CLINICAL TRIAL: NCT06780943
Title: Quantification of Motor Compensation Following Biomechanical, Proprioceptive and Physiological Alterations Post-lower Limb Amputation.
Acronym: QAMPA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2024/EP-02
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Amputation
MeSH Terms: interventions — Biomechanical Phenomena

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Transtibial amputee patients
  Interventions: Other: Biomechanics; Other: Physiological; Other: Proprioceptive
- Transfemoral amputee patients
  Interventions: Other: Biomechanics; Other: Physiological; Other: Proprioceptive
- Healthy volunteers
  Interventions: Other: Biomechanics; Other: Physiological; Other: Proprioceptive

INTERVENTIONS:
Other: Biomechanics — Amputees and controls will be equipped with measurement sensors to record spatio-temporal, kinetic, kinematic, pressure, electromyographic and physiological parameters of gait in the movement analysis laboratory (GRAIL System).
  16 Anatolog FSR sensors will be installed in the amputee population (transtibial, transfemoral on the medial, lateral, anterior and posterior parts of the stump, 4 per side, aligned in the proximal/distal axis. The Anatolog sensors have a sampling frequency of 100Hz. Electromyographic data recording is performed by setting up a number of EMGs depending on the healthy population or the level of amputation. Surface electromyography (sEMG) signals will be recorded from 10 muscles on each lower limb for control subjects and transtibial amputees
Other: Physiological — Energy consumption (VO2), will be performed using the VO2 Master Pro (VO2 Master Health Sensors Inc., Vernon, British Columbia, CA). Each participant will wear a face mask connected to the VO2 Master, which will measure oxygen consumption in real time during the assessment. The mask will be adjusted to prevent air leakage and ensure accurate measurements.
Other: Proprioceptive — For amputees, the joint above the amputation will be measured due to the presence of the proximal insertions of the bi-articular muscles and the absence of their distal insertion (i.e., knee joint for transtibial amputees and hip joint for transfemoral amputees).

SUMMARY:
Lower limb amputation causes segmental loss that alters locomotor organization. The human body, designed to function in a multisegmental manner, must adapt to this new configuration where segments are missing, depending on the level of amputation. These adaptations are directly linked to the biomechanical, physiological and proprioceptive alterations caused by the loss of the amputated segments. Without mechanoreceptive afferents essential for regulating locomotion, the sensory system uses alternative information to maintain efficient locomotor function. The prosthesis partially compensates, but remains limited on the biomechanical and proprioceptive levels. Current prosthetic technologies, inspired by biomimicry, aim to imitate evolutionary solutions to restore walking, although current algorithms do not allow real-time modulation. This research aims to characterize post-amputation locomotor adaptations through biomechanical, physiological and proprioceptive exploration to develop a "locomotor characterization" model.

The study authors hypothesize that the post-amputation alterations are exacerbated in contexts of continuous and discontinuous constraints (e.g., ascent/descent and destabilization), and that the addition of a prosthesis, although inspired by biomimicry, only restores partial compensation of locomotor functions.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Persons with unilateral transtibial or transfemoral amputees followed in the MPR department at the Nîmes University Hospital, RRL department, Grau du Roi University Rehabilitation Hospital.
* All etiologies: vascular, traumatic and septic.
* Adapted equipment validated by the rehabilitation doctor.
* Able to walk for 5 minutes on a treadmill without technical assistance

Inclusion criteria specific to healthy volunteers:

* Adults (>18 years old) and under 40 years old
* Able to walk for 5 minutes on a treadmill without technical assistance.
* Body mass index between 18 and 25

Exclusion Criteria:

* The patient is participating in an interventional or a drug/medical device study, or is in a period of exclusion determined by a previous study
* The patient unable to express consent
* It is impossible to give the patient informed information
* The patient is under safeguard of justice or state guardianship
* Patient who has already been included in this study.
* Pregnant, parturient or breastfeeding patient.
* Appearance of a stump wound during the study requiring unloading.
* Patient for whom the implementation of vibration stimulation is not possible

Exclusion criteria for amputee patients:

* Patient suffering from uncorrected or untreated visual disorders.
* Patient with major cognitive disorders (MoCA <23).
* Patient with vestibular disorders or uncontrolled epilepsy.
* Patient with an unhealed amputation stump.
* Patient with a weight > 135kg or < 20kg
* Patients with a FAC of 1 (i.e. patients who need firm and continuous assistance from a person to support their weight and maintain balance) or less.
* Sensory impairment that makes it impossible to perceive stimulation
* Significantly reduced bone density
* Patient in whom it is impossible to correctly adjust the GRAIL System harness to the corresponding body part due to:

  * Body shape
  * Colostomy bags
  * Skin lesions that cannot be adequately protected.
  * Any other reason that prevents a good, painless adjustment of the harness.
* Patient in whom it is impossible to correctly adjust the CON-TREX System:

  * Body shape
  * Colostomy bags
  * Skin lesions that cannot be adequately protected.
  * Any other reason that prevents a good, painless adjustment of the support systems.

Exclusion criteria for healthy volunteers:

* History of significant injury or surgery affecting the lower limbs (such as hip or knee replacement or knee/ankle ligament reconstruction) that could impact walking
* History of neurological or psychiatric disorders that could affect locomotion or the processing of sensorimotor information.
* Drug treatments affecting locomotion: drugs likely to alter walking or balance, such as sedatives, muscle relaxants or neuroleptics.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Person with unilateral transtibial or transfemoral amputation and healthy volunteers for control population.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Locomotor adaptations induced by amputations on inter-segmental coordination by the evaluation of continuous relative phases under different walking conditions | Day 0
  MARP (Mean Absolute Relative Phase) index of Continuous Relative Phases (movement analysis) where MARP = 0 indicates perfectly synchronization in both segments throughout the gait cycle and elevated MARP indicates poor coordination between the segments

SECONDARY OUTCOMES:
Locomotor adaptations induced by amputations on the impact of locomotor constraints such as inclinations on the explanation of muscular synergies under different walking conditions | Day 0
  Muscle synergy explanation index
Locomotor adaptations induced by amputations on the extent of locomotor constraints such as inclinations on the explanation of muscular synergies under different walking conditions | Day 0
  Number of muscle synergies
Locomotor adaptations induced by amputations on the variability of pressure distributions in the socket under different walking conditions | Day 0
  Variability of pressures in the socket measured with high-pressure Force-Sensing Resistor sensor. The variability will be determined according to the standard deviation of all 16 pressures measured during a walking cycle.
Locomotor adaptations induced by amputations on oxygen consumption under different walking conditions | Day 0
  Average VO2 in the final 30 seconds of walking (mL/mn/kg)
Locomotor adaptations induced by amputations on energy consumption under different walking conditions | Day 0
  Cost of the task defined by the difference in O2 consumption during walking compared to O2 consumption at rest.
Locomotor adaptations induced by amputations on heart rate under different walking conditions | Day 0
  Beats per minute
Characterize the proprioceptive deficits induced by amputations on the angular precision of the joints | Day 0
  Reduction of the angular matching error, where the unilateral angular positioning error is measured as the difference in angular data between the reference angle and the estimated angle
Characterize the proprioceptive deficits induced by amputations on movement perception | Day 0
  Angular displacement detection threshold (°)
Characterize the proprioceptive deficits induced by amputations on response time | Day 0
  Response time for angular matching (ms)
Characterize the proprioceptive deficits induced by amputations on angular displacement | Day 0
  Angular displacement direction detection (%)
Identify a method for restoring proprioceptive deficits via modulation of the "optimal" frequency and amplitude | Day 0
  Proprioception index (average of the different errors and detection thresholds)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Pantera, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No